CLINICAL TRIAL: NCT05551611
Title: Vaginal Breech Birth Management Educational Mobile Game Design and Evaluation for Midwifery Students
Brief Title: Vaginal Breech Birth Management Educational Mobile Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: Kocaeli University (Other); Marmara University (Other)
Responsible Party: Principal Investigator, Suzi Özdemir, Investigator, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Suzi-01
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Vaginal Breech Delivery Management; Mobile Game
Keywords: Midwifery; mobile game; vaginal breech delivery management; midwifery education
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Playgroup (Active Comparator): The participants were informed about the research and the mean score was calculated by applying the Vaginal Breech Delivery Management Knowledge Test to the participants before the vaginal delivery management training of the breech-presented fetus was given within the scope of the Risky Delivery and Postpartum Period Course. After playing the mobile game, Vaginal Breech Birth Management Post-Knowledge Test and General Satisfaction Level Test were applied to the participants again. In addition, the Mobile Game Evaluation Form was applied to the participants in the game group and their opinions on the mobile educational game were determined. Test-retest reliability was calculated by applying the Vaginal Breech Delivery Management Knowledge Retention Test 14 days later.
  Interventions: Other: Playgroup
- Control group (Active Comparator): The participants were informed about the research and the mean score was calculated by applying the Vaginal Breech Delivery Management Knowledge Test to the participants before the vaginal delivery management training of the breech-presented fetus was given within the scope of the Risky Delivery and Postpartum Period Course. On the same date as the playgroup, but at a different time and in a class, the researcher gave a theoretical lesson through the presentation prepared in the powerpoint program about the birth management of a breech-presented fetus in the classroom as in the traditional education method. After the lesson, the Vaginal Breech Birth Management Post-Knowledge Test and the General Satisfaction Level Test were administered to the participants again. Test-retest reliability was calculated by applying the Vaginal Breech Delivery Management Knowledge Retention Test 14 days later.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Playgroup — The mobile game will be sent to the students via a link and the students are allowed to install it on their mobile phones with android and ios operating systems. The internet required for the download was provided by the researcher. For the students who did not have a smart phone in the playgroup, the game would be started from the researcher's phone and the game was played sequentially. All students were allowed to use headphones while playing the game. In order to log in to the game, an account was created on behalf of each student, and the game user name and password were sent to the students by e-mail. It was ensured that they did not communicate with anyone and did not receive help during the game with the supervision of the researcher. Waited until each participant completed the game. Then, the mobile game was deleted from the smartphones of all participants, and the download link was inactive until the research process was completed.
  Arms: Playgroup
Other: Control group — The researcher gave a theoretical lesson through the presentation prepared in the powerpoint program about the birth management of a breech-presented fetus in the classroom as in the traditional education method.
  Arms: Control group

SUMMARY:
Mobile games are used as a powerful learning tool today. It is very useful as it allows students to work on their own frequently when necessary without the need for any physical environment or trainer and can be easily distributed among institutions. While the simulation laboratories established in a school can only be used by the students of that school, a game developed can be used by all students in the world who know that language.

It is reported that breech presentation, which is one of the presentation disorders of the fetus, is the fourth or fifth most common indication for delivery by cesarean section. According to the midwifery national core curriculum in our country, vaginal breech delivery management training is given within the scope of risky birth course. However, it is known that teaching and learning the labor and delivery process of a breech-presented fetus is not easy. For this reason, it is thought that teaching vaginal breech delivery management by gamifying will be beneficial and it is important to investigate the effect of students playing this game on learning.

Our study has two aims. Its primary purpose is; is to design a vaginal breech delivery management educational mobile game for midwifery students. The secondary aim is to evaluate the effect of the educational mobile game-supported teaching activity given to midwifery students about vaginal breech delivery within the scope of risky birth and postpartum period course.

Real actors and simulation models were used to fake the scenario to be used in the game. A mobile game was prepared with the film shot. It was conducted with 10 volunteer students from Marmara University Health Sciences Faculty Midwifery Department 3rd grade students in order to determine whether there is any aspect of the mobile game that requires development. The mobile game, which was shaped and organized with the pilot application, was applied to the students in the 3rd grade play group of Kocaeli University Health Sciences Faculty Midwifery Department after single-blind randomization. Introductory features form, vaginal breech birth management knowledge test, course effectiveness evaluation form, general satisfaction level test about the course and vaginal breech birth management mobile game evaluation form were used to collect data.

DETAILED DESCRIPTION:
H1: There is a statistically significant difference between the Vaginal Breech Birth Management Post-Test of Knowledge scores of the students in the play group and the students in the control group.

H2: There is no statistically significant difference between the mean scores of the students in the play group and the students in the control group in the Vaginal Breech Birth Management Post-Test of Knowledge.

H3: There is a statistically significant difference between the Vaginal Breech Birth Management Knowledge Retention Test mean scores of the students in the play group and the students in the control group.

H4: There is no statistically significant difference between the Vaginal Breech Birth Management Knowledge Retention Test mean scores of the students in the play group and the students in the control group.

Variables of the Study Independent variable Playing the vaginal breech delivery management mobile game for the students taking the Normal Birth and Postpartum Period course The dependent variable Vaginal breech birth management knowledge test, course effectiveness evaluation form, general satisfaction level test for the course, mobile game evaluation forms Research Design It is a prospective, single-blind, randomized controlled experimental type study with a pretest-posttest design.

Place and Time of Research The research is carried out with 3rd grade students within the scope of Risky Birth and Postpartum Term course in the 2021-2022 academic year spring semester at Kocaeli University, Faculty of Health Sciences, Midwifery Department, and the pilot application of the research is carried out with 3rd grade students of the Midwifery Department of Marmara University Health Sciences Faculty.

Population and Sample of the Research The universe of the research consists of 81 3rd grade midwifery students from Kocaeli University Faculty of Health Sciences in the 2021-2022 academic year in order to be the institution where the researcher works and to facilitate data collection. According to the sample calculation, it was planned to reach at least 68 students at the 5% Type 1 error level and the 95% confidence interval. It was planned to apply the study to the whole population in order to prevent possible case losses. A total of 79 students were included in the sample because two of the students did not attend the classes.

Ethical aspect of research Ethics committee approval for the study was received from Kocaeli University Non-Interventional Clinical Research Ethics Committee (approval date / decision no: GOKAEK-2022/02.11) on 28.01.2022. Written permissions were obtained from the Kocaeli University Faculty of Medicine Dean's Office for the use of the simulation laboratory, where the scenario will be filmed, from the Marmara University Faculty of Health Sciences for the pilot application of the play, and from the Kocaeli University Faculty of Health Sciences Dean's Office for the implementation phase of the study. During the preliminary and pilot implementation, the participants were informed verbally and in writing about the purpose of the research and that their personal information would be kept confidential. However, it was stated to the participants that participation in the study was on a voluntary basis and if they submitted the study forms, they would be deemed to have given their consent to participate in the study. Our study is carried out in accordance with the Principles of the Declaration of Helsinki.

Randomization and creation of groups Kocaeli University Faculty of Health Sciences, 2021-2022 academic year, 81 3rd grade midwifery students were divided into experimental and control groups using the computer-assisted (www.randomizer.org) randomization program. The experimental group was called the play group, and the other group was called the control group.

All students will be asked not to share their intervention experiences until the research process is completed by the researcher.

During the research process, the traditional education method will not be explained to the students in the play group and the delivery management of the breech-presented fetus, and the vaginal breech delivery management mobile game will not be played to the students in the control group. After the study process is completed, both education methods will be applied to the students in both groups.

Development of the Mobile Game to be Used in the Research In the prepared mobile game, the labor process of the pregnant was recorded with the actors acting, and the breech birth scene was recorded using simulation models.

The creation of mobile game content consists of five parts. In the first part, the determination of the game to be digitized and the creation of the game-specific scenario and scenario questions are included, while the second part includes the presentation of the scenario and scenario questions to expert opinions. In the third part, the film is shot by putting the scenario on the stage, and the transfer of the film shot in the fourth part to the mobile game and the pilot application of the game are included. In the fifth section, which is the last section, the effectiveness of the vaginal breech delivery management mobile game developed on the 3rd grade students of the Department of Midwifery, Faculty of Health Sciences, Kocaeli University, was evaluated.

First part: The story of the game, characters related to the game and questions about the player were created in line with the relevant literature in determining the game and creating the original scenario.

Second part: The scenario and scenario questions were sent to eight academicians who are experts in the field of midwifery and have at least five years of academic experience, and seven clinician midwives with at least five years of delivery room experience. Areas were created to evaluate the submitted scenario as positive and negative for each section's features, and experts were asked to express their views on those areas. In line with the evaluations received, the final version of the scenario and scenario questions were obtained. The draft of the script was then scripted by a screenwriter and the lines were created.

Third part: Real actors and simulation models were used to fake the script. Film and model simulation shooting was carried out with a professional team at Kocaeli University Good Physician Practices and Simulation Center, where the necessary institutional permission was obtained, with the role of professional actors, whose consent was obtained before. The creation of realistic scenes was provided by the necessary equipment (make-up, professional camera, etc.).

Pregnant and her partner were played by two professional actors. A fake pregnant belly model was applied to the woman who assumed the role of pregnant with the help of professional make-up. In applications performed from the abdominal region such as the Leopold maneuver, electronic fetal monitoring application, and FKA listening, the abdomen of the pregnant woman was opened so that only the abdominal region was visible. In midwifery practices such as vaginal examination, no demonstration was made, but the impression that vaginal examination would be performed was reflected. During the movie, a gimbal camera was used at the head of the actor who will play the role of a midwife. In this way, it was ensured that the event pattern was observed from the eyes of the midwife.

During the birth, the moment of birth was animated with models by using simulation models. The camera is set to record only maneuvers used at the time of birth and postpartum procedures.

The fourth part: In the transfer of the film to the mobile game, individual service was received from an information system engineer who is an expert in his field.

In the mobile game, questions appear on the screen at certain intervals during the movie, and the movie continues to play after the student answers the question. When the student gives a wrong answer to the question, a text is displayed stating why that answer is wrong. In cases where filming was appropriate, the results of the wrong choice were transferred to the film and the actor was able to visually and audibly watch the result of the wrong answer. Playing the game takes an average of 30-45 minutes.

In order for students to access the mobile game, a different user name and password were created for each student. The link required to download the game and the username and password that were created before to enter the game were sent to the student by the researcher over the internet (e-mail/WhatsApp).

After the game was developed, a pilot application was made. This app helped determine how long it would take to complete the mobile game and whether there were any aspects of the game that needed improvement. The pilot application of the game and measurement tools was carried out with 10 volunteer students from the 3rd grade students of the Department of Midwifery, Faculty of Health Sciences, Marmara University, for which the necessary institutional permission was obtained.

Fifth Part: The mobile game, which was shaped and organized with the pilot application, was applied to the students in the 3rd grade playgroup of Kocaeli University Faculty of Health Sciences Midwifery Department after single-blind randomization on May 13, 2022.

Data Collection Forms Introductory features form, vaginal breech birth management knowledge test, course effectiveness evaluation form, general satisfaction level test for the course, vaginal breech birth management mobile game evaluation forms were used to collect data. All forms to be used in data collection were submitted to expert opinions after obtaining ethical committee permission and institutional permissions, and they were finalized.

Introductory features form: It is the form in which the socio-demographic and previous knowledge of digital game playing of the students participating in the study are questioned.

Vaginal breech birth management knowledge test: A questionnaire was created in line with the relevant literature in line with the content of the risky birth and postpartum course in order to provide the necessary knowledge and skills for the management of the labor and delivery process of the pregnant with the fetus in breech presentation, to make appropriate interventions, and to adopt the roles and responsibilities of the midwife. The created questionnaire was presented to the expert opinion along with the scenario, and it was finalized in line with the feedback received. These questions will be evaluated with the assessment and evaluation system developed independently of the educational mobile game. Each correct answer is 1 point, and the maximum score that can be obtained from the test will be determined by the number of questions.

Course effectiveness evaluation form: The form, which was prepared by the researchers in line with the literature review, was applied to the play group after the vaginal breech delivery management mobile game was played, and to the control group after the birth management training of the breech presentation fetus, which was given through traditional education. In this questionnaire, there are statements that allow the evaluation of the education given by the student. The minimum score to be taken from the form to be evaluated with a 5-point Likert-type (1=Totally disagree, 2=Disagree, 3=Undecided, 4=Agree, 5=Totally Agree) is 11, and the maximum score is 55.

General satisfaction level test for the lesson: It was applied to the play group after the vaginal breech management educational mobile game was played, and to the control group after the birth management training of the breech presentation fetus, which was given through traditional education. The test, in which the participants will be asked to indicate their general level of satisfaction with the lesson, will be evaluated with a 6-point Likert type, and the average score of the test in both groups was calculated.

Vaginal breech delivery management mobile game evaluation form: It is a questionnaire developed by the researchers in line with the literature review to evaluate the clarity and convenience, suitability and quality of the mobile game by the players. In this survey; The harmony of the text, fonts and colors of the game, the legibility of the size and style, the attractiveness and clarity of the game design (interface, graphics, etc.), the ease of learning and playing, the state of the game's content and structure to increase the player's knowledge and self-confidence about the subject, the fluency of the game, the lesson. There are expressions that evaluate the opinions of the players, such as the situation of being a reinforcing tool. The minimum score to be taken from the form to be evaluated with a 5-point Likert type (1=I totally disagree, 2=Disagree, 3=Undecided, 4=Agree, 5=Completely Agree) is 39, and the maximum score is 195.

Statistical analysis will be performed using the IBM SPSS Statistic 22.0 (IBM Corp., Armonk, NY, USA) program. Descriptive statistical methods (number, percentage, mean, standard deviation) will be used in the evaluation of socio-demographic data. Parametric tests (chi-square, T test, etc.) will be used in the comparison of categorical variables when the data are found to be suitable for normal distribution, and non-paramedic tests (Mann-Whitney U Test, Kruskal Wallis, etc.) will be used when they are not suitable for normal distribution.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Being a midwifery student,
* Being a 3rd year student at Kocaeli University, Faculty of Health Sciences, Department of Midwifery,
* To have taken the Normal Birth and Postpartum Period course.

Exclusion Criteria:

* Not having a mobile phone or using mobile games
* Leaving the research process for any reason
* To have received practical or theoretical training on breech birth before
* Being unable to speak, read and write Turkish

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Özlem Çağan, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Play Group: The participants were informed about the research and the mean score was calculated by applying the VBBM Knowledge Test to the participants before the vaginal delivery management training of the breech-presented fetus was given within the scope of the Risky Delivery and Postpartum Period Course. After playing the mobile game, VBBM Post-Knowledge Test and General Satisfaction Level Test were applied to the participants again. In addition, the Mobile Game Evaluation Form was applied to the participants in the game group and their opinions on the mobile educational game were determined. Test-retest reliability was calculated by applying the Vaginal Breech Delivery Management Knowledge Retention Test 14 days later.
Period: Overall Study
Arm/Group | Play Group | Control Group
Started | 39 | 40
Completed | 39 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: SPSS 23 program was used for data analysis.
Groups:
- Playgroup: The participants were informed about the research and the mean score was calculated by applying the VBBM Knowledge Test to the participants before the vaginal delivery management training of the breech-presented fetus was given within the scope of the Risky Delivery and Postpartum Period Course. After playing the mobile game, VBBM Post-Knowledge Test and General Satisfaction Level Test were applied to the participants again. In addition, the Mobile Game Evaluation Form was applied to the participants in the game group and their opinions on the mobile educational game were determined. Test-retest reliability was calculated by applying the Vaginal Breech Delivery Management Knowledge Retention Test 14 days later.
- Control Group: The participants were informed about the research and the mean score was calculated by applying the VBBM Knowledge Test to the participants before the vaginal delivery management training of the breech-presented fetus was given within the scope of the Risky Delivery and Postpartum Period Course. On the same date as the playgroup, but at a different time and in a class, the researcher gave a theoretical lesson through the presentation prepared in the powerpoint program about the birth management of a breech-presented fetus in the classroom as in the traditional education method. After the lesson, the VBBM Post-Knowledge Test and the General Satisfaction Level Test were administered to the participants again. Test-retest reliability was calculated by applying the Vaginal Breech Delivery Management Knowledge Retention Test 14 days later.
- Total: Total of all reporting groups
Arm/Group | Playgroup | Control Group | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.15 (0.84) | 21.13 (0.85) | 21.14 (0.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 79
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 39 | 40 | 79
Vaginal Breech Birth Management Knowledge Test [Median (Inter-Quartile Range); unit: units on a scale] — A 52-item questionnaire on midwives' breech birth knowledge was developed and reviewed by 12 experts, showing high content validity (CVI=0.98) and strong agreement (Kendall's W=0.70; p<0.001). Based on feedback, two items were removed, and ten were revised. A pilot test with 10 students confirmed clarity. Internal consistency (KR-20) was 0.612 after removing three items, showing acceptable reliability. Scores range from 0 to 47, with higher scores indicating better knowledge. The finalized questionnaire was given to experimental and control groups at specified intervals.
  units on a scale | 36 [34 to 40] | 35 [31.25 to 38.75] | 35.5 [32.62 to 39.37]

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Effectiveness of Vaginal Breech Birth Management Serious Mobile Game
Description: The Vaginal Breech Birth Management Knowledge Test (VBBM-KT) is a 47-item multiple-choice assessment developed to evaluate midwifery students' knowledge of vaginal breech birth trauma and management.
  * Each correct answer scores 1 point, resulting in a total score range from 0 to 47 points.
  * There are no subscales; only a total score is calculated.
  * Higher scores represent better knowledge and indicate a more successful learning outcome.
  The test was administered to both groups at four time points: pre-intervention (pretest), immediately post-intervention (Day 0), two weeks later (Day 14), and seven months later.
Time Frame: Pretest, posttest (Day 0), 14 days after intervention (14th day), and 7 months after intervention (7th month)
Population: The sample group consists of all third-year midwifery students.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Playgroup: A serious mobile game was used to teach vaginal breech birth management.
- Control Group: Traditional teaching method have been used for teach vaginal breech birth management.
Arm/Group | Playgroup | Control Group
Number analyzed (Participants) | 39 | 40
units on a scale
  vaginal breech birth management knowledge test (pretest) | 36.51 (3.26) | 34.75 (4.98)
  vaginal breech birth management knowledge test (posttest) | 40.46 (4.21) | 37.77 (5.12)
  vaginal breech birth management knowledge test (14th day) | 38.00 (4.08) | 37.05 (3.77)
  vaginal breech birth management knowledge test (7th month) | 35.48 (3.78) | 35.77 (5.07)

ADVERSE EVENTS:
Time Frame: 7 months
Description: The mobile game or narrative method may cause discomfort and frustration for participants due to prolonged sitting, improper operation of the device or distraction.
Arm/Group | Playgroup | Control Group
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 0/39 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT05551611/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT05551611/ICF_001.pdf